CLINICAL TRIAL: NCT02859350
Title: Age Escalation / De-escalation Study to Evaluate the Safety, Tolerability and Immunogenicity of a Radiation-attenuated Plasmodium Falciparum (Pf) Sporozoite Vaccine (PfSPZ Vaccine) in Equatoguinean Adults, Children and Infants, and Comparison With Non-attenuated Pf Sporozoites (PfSPZ Challenge) Administered Under Chloroquine Prophylaxis (PfSPZ-CVac Approach) for Efficacy Against Controlled Human Malaria Infection.
Brief Title: Safety, Tolerability and Immunogenicity of PfSPZ Vaccine in an Age De-escalation Trial in Equatorial Guinea.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Ifakara Health Institute (Other); Swiss Tropical & Public Health Institute (Other); Government of Equatorial Guinea (Other Government); Marathon Oil Corporation (Industry); Noble Oil Services (Industry); La Paz Medical Center, Malabo, Equatorial Guinea (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EGSPZV2
Record Dates: First submitted 2016-07-27; First posted 2016-08-09 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; PfSPZ Vaccine; PfSPZ Challenge (NF54); CHMI; Chloroquine; Chemoprophylaxis; PfSPZ-CVac
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (15):
- Group 1a (PfSPZ Vaccine) (Experimental): 18-35 years; n= 20; 3 doses of 2.7x10^6 PfSPZ Vaccine given eight weeks apart. Volunteers will receive CHMI between 10 and 14 weeks post last vaccination (with a window of +/-7 days on each side) and will be followed for 8 weeks following CHMI.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (for CHMI)
- Group 1a (normal saline) (Placebo Comparator): 18-35 years; n=6; 3 doses of normal saline given 8 weeks apart. Volunteers will receive CHMI between 10 and 14 weeks post last dose of NS (with a window of +/-7 days on each side) and will be followed for 8 weeks following CHMI.
  Interventions: Biological: PfSPZ Challenge (for CHMI); Other: Normal Saline
- Group 1b (PfSPZ CVac) (Experimental): 18-35 years; n=20; 3 doses of 1.0x10^5 PfSPZ Challenge given every four weeks. Group 1b will start 8 weeks after Group 1a. Volunteers in Group 1b will receive their first immunization after the loading dose of chloroquine has been administered. Volunteers will receive CHMI between 10 and 14 weeks post last vaccination (with a window of +/-7 days on each side) and will be followed for 8 weeks following CHMI.
  Interventions: Biological: PfSPZ Challenge (for CHMI); Biological: PfSPZ Challenge (for PfSPZ-CVac)
- Group 1b (normal saline) (Placebo Comparator): 18-35 years; n=6; 3 doses of normal saline given 4 weeks apart. Group 1b will start 8 weeks after Group 1a. Volunteers will receive CHMI between 10 and 14 weeks post last dose of NS (with a window of +/-7 days on each side) and will be followed for 8 weeks following CHMI.
  Interventions: Biological: PfSPZ Challenge (for CHMI); Other: Normal Saline
- Group 2 (PfSPZ Vaccine) (Experimental): 36-65 years; n=12; 3 doses of 2.7x10^6 PfSPZ Vaccine given 8 weeks apart. Group 2 will start 3 weeks after Group 1a.
  Interventions: Biological: PfSPZ Vaccine
- Group 2 (normal saline) (Placebo Comparator): 36-65 years; n=4; 3 doses of normal saline given 8 weeks apart. Group 2 will start 3 weeks after Group 1a.
  Interventions: Other: Normal Saline
- Group 3 (PfSPZ Vaccine) (Experimental): 11-17 years; n=12; 3 doses of 1.8x10^6 PfSPZ Vaccine given 8 weeks apart. Group 3 will start 3 weeks after Group 1a.
  Interventions: Biological: PfSPZ Vaccine
- Group 3 (normal saline) (Placebo Comparator): 11-17 years; n=4; 3 doses of normal saline given 8 weeks apart. Group 3 will start 3 weeks after Group 1a.
  Interventions: Other: Normal Saline
- Group 4 (PfSPZ Vaccine) (Experimental): 6-10 years; n=12; 3 doses of 1.8x10^6 PfSPZ Vaccine given 8 weeks apart. Group 4 will start 4 weeks after Group 1a.
  Interventions: Biological: PfSPZ Vaccine
- Group 4 (normal saline) (Placebo Comparator): 6-10 years; n=4; 3 doses of normal saline given 8 weeks apart. Group 4 will start 4 weeks after Group 1a.
  Interventions: Other: Normal Saline
- Group 5 (PfSPZ Vaccine) (Experimental): 1-5 years; n=12; 3 doses of 1.8x10^6 PfSPZ Vaccine given 8 weeks apart. Group 5 will start 7 weeks after Group 1a.
  Interventions: Biological: PfSPZ Vaccine
- Group 5 (normal saline) (Placebo Comparator): 1-5 years; n=4; 3 doses of normal saline given 8 weeks apart. Group 5 will start 7 weeks after Group 1a.
  Interventions: Other: Normal Saline
- Group 6a (PfSPZ Vaccine) (Experimental): 6-11 months; n=3; 1 dose of 9.0x10^5 PfSPZ Vaccine. Group 6a will start 7 weeks after Group 1a.
  Interventions: Biological: PfSPZ Vaccine
- Group 6b (PfSPZ Vaccine) (Experimental): 6-11 months; n=12; 3 doses of 1.8x10^6 PfSPZ Vaccine given 8 weeks apart. Group 6b will start 11 weeks after Group 1a.
  Interventions: Biological: PfSPZ Vaccine
- Group 6b (normal saline) (Placebo Comparator): 6-11 months; n=4; 3 doses of normal saline given 8 weeks apart. Group 6b will start 11 weeks after Group 1a.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: PfSPZ Vaccine — Metabolically active, non-replicating, radiation attenuated, aseptic, purified, cryopreserved NF54 P. falciparum (Pf) sporozoites (PfSPZ Vaccine)
  Arms: Group 1a (PfSPZ Vaccine); Group 2 (PfSPZ Vaccine); Group 3 (PfSPZ Vaccine); Group 4 (PfSPZ Vaccine); Group 5 (PfSPZ Vaccine); Group 6a (PfSPZ Vaccine); Group 6b (PfSPZ Vaccine)
Biological: PfSPZ Challenge (for CHMI) — live, infectious, aseptic, purified, cryopreserved NF54 P. falciparum (Pf) sporozoites (PfSPZ Challenge) Controlled human malaria infection (CHMI) by direct venous inoculation of 3,200 PfSPZ Challenge
  Arms: Group 1a (PfSPZ Vaccine); Group 1a (normal saline); Group 1b (PfSPZ CVac); Group 1b (normal saline)
Other: Normal Saline — 0.9% Sodium chloride
  Arms: Group 1a (normal saline); Group 1b (normal saline); Group 2 (normal saline); Group 3 (normal saline); Group 4 (normal saline); Group 5 (normal saline); Group 6b (normal saline)
Biological: PfSPZ Challenge (for PfSPZ-CVac) — live, infectious, aseptic, purified, cryopreserved NF54 P. falciparum (Pf) sporozoites (PfSPZ Challenge)
  Arms: Group 1b (PfSPZ CVac)

SUMMARY:
This trial will evaluate the safety, tolerability, and immunogenicity of PfSPZ Vaccine in healthy Equatoguinean adults, adolescents, children and infants who receive doses of 0.9x10^6, 1.8x10^6 or 2.7x10^6 PfSPZ Vaccine via direct venous inoculation (DVI) compared with control groups receiving normal saline (NS) placebo by DVI. In addition, the study will also assess a second PfSPZ-based vaccination approach known as PfSPZ-CVac- the administration of non-irradiated, infectious PfSPZ (PfSPZ Challenge) (1x10^5 PfSPZ) under anti-malarial chemoprophylaxis (chloroquine) in younger adults ages 18 to 35 years for safety, tolerability, immunogenicity and efficacy against controlled human malaria infection (CHMI).

DETAILED DESCRIPTION:
EGSPZV2 is a single center, double-blind, placebo-controlled trial. The study is to take place at the Baney Temporary Research Facility (BTRF) located in Baney City. One hundred and thirty-five healthy male and female; adults, adolescents, children and infant volunteers, aged from 6 months to 65 years who live in the Baney district and Malabo city on Bioko Island will be enrolled based on pre-defined inclusion and exclusion criteria implemented according to international ethical standards.

The trial will consist of seven groups (Group 1a: younger adults, ages 18-35; Group 2: older adults, ages 36-65; Group 3: adolescents, ages 11-17; Group 4: older children, ages 6-10; Group 5: younger children, ages 1-5; Groups 6a/b: infants, ages 6 months - 11 months) of volunteers. Vaccination will begin in Group 1a (younger adults), with three doses of 2.7x10^6 PfSPZ Vaccine given eight weeks apart by DVI. An eighth group (Group 1b: younger adults, ages 18- 35), will be uniquely immunized with the comparator vaccine PfSPZ Challenge given under chloroquine prophylaxis (PfSPZ-CVac approach), rather than with PfSPZ Vaccine. A single PfSPZ-CVac younger adult group (group 1b) is included to provide a direct comparison with PfSPZ Vaccine (group 1a) for the ability to protect against CHMI. Each of the first two groups (1a and 1b) will have 20 participants receiving either PfSPZ Vaccine or PfSPZ Challenge and 6 participants receiving NS placebo by DVI, with treatment allocation randomized and double-blind. Volunteers in Group 1b will receive vaccinations 8 weeks after the initial vaccination of Group 1a. Volunteers in Group 1 (younger adults) will receive CHMI between 10 and 14 weeks post last vaccination (with a window of +/- 7 days on each side) and will be followed for 8 weeks following CHMI.

Group 2 (older adults) will receive three doses of 2.7x10^6 PfSPZ Vaccine. Group 2 will consist of 12 participants receiving PfSPZ Vaccine and 4 participants receiving NS placebo by DVI, given eight weeks apart. Group 3, 4, 5 and 6b will each have 12 participants receiving three doses of 1.8x10^6 PfSPZ Vaccine and 4 participants receiving NS, also given eight weeks apart. Group 6a will consist of 3 volunteers who will receive a single dose of 9.0 x10^5 PfSPZ Vaccine.

Sequential age groups will be staggered to allow assessment of safety and tolerability before further age de-escalation. To assure safety, vaccinations will start in younger adults and will progress to younger and older age groups using staggered start dates at approximately weekly intervals. Age escalation and initial age de-escalation will take place at the same time, hence Group 2 and 3 will be vaccinated at the same time. Progressively younger age groups will then be immunized. The decision to proceed with each of these steps will be made by the study team after a review of safety data from the previously vaccinated group(s). Three Safety Monitoring Committee (SMC) meetings are scheduled to review data prior to initiating the younger children and infant groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, based on clinical and laboratory findings
* From the age 6 months to 65 years
* Adults with a Body Mass Index (BMI) 18 to 30 Kg/m2; or adolescents, children and infants with Z-score of the selected indicator ([weight-for-height], [(height and BMI) for age]) category within ±2SD as detailed in protocol
* Long-term (at least one year) or permanent residence in the Baney district or Malabo city
* Agreement to release medical information and to inform the study doctor concerning contraindications for participation in the study
* Willingness to be attended to by a study clinician and take all necessary medications prescribed during study period
* Agreement to provide contact information of a third party household member or close friend to study team
* Agreement not to participate in another clinical trial during the study period
* Agreement not to donate blood during the study period
* Able and willing to complete the study visit schedule over the study follow up period, including the hospitalizations required for protocol compliance
* .Willingness to undergo HIV, hepatitis B (HBV) and hepatitis C (HCV) tests
* Volunteer (subjects 18 years of age and older) or the parent / guardian signing the informed consent (for subjects <18 years of age) is able to demonstrate their understanding of the study by responding correctly to 10 out of 10 true/false statements (in a maximum of two attempts for those who failed to respond correctly to all true/false statements in the first attempt).
* Signed written informed consent, in accordance with local practice, provided by adult volunteers, parents or legal representatives and relevant assent for children participants as applicable.
* Free from malaria parasitemia by blood smear at enrollment and by PCR for group 1
* Has not been treated with any antimalarial medication for at least two weeks prior to the first immunization.
* Free from helminth infections (detected by microscopy) at enrollment.
* Female volunteers aged 9 years and above must be non-pregnant (as demonstrated by a negative urine pregnancy test), and provide consent/assent of their willingness to take protocol-defined measures not to become pregnant during the study and safety follow-up period.

Exclusion Criteria:

* Previous receipt of an investigational malaria vaccine in the last 5 years
* Participation in any other clinical study involving investigational medicinal products including investigational malaria drugs within 30 days prior to the onset of the study or during the study period
* History of arrhythmias or prolonged QT-interval or other cardiac disease, or clinically significant abnormalities in electrocardiogram (ECG) at screening
* Positive family history in a 1st or 2nd degree relative for cardiac disease at age <50 years old
* A history of psychiatric disease
* Suffering from any chronic illness including; diabetes mellitus, cancer or HIV/AIDS
* Any confirmed or suspected immunosuppressive or immune-deficient condition, including asplenia
* History of drug or alcohol abuse interfering with normal social function
* The use of chronic immunosuppressive drugs or other immune modifying drugs within three months of study onset (inhaled and topical corticosteroids are allowed) and during the study period
* Any clinically significant deviation from the normal range in biochemistry or hematology blood tests or in urine analysis
* Positive HIV, hepatitis B virus or hepatitis C virus tests
* Volunteers who are have risk factors for tuberculosis and/or signs and symptoms of tuberculosis (TB), plus a positive tuberculin skin test (TST).
* Symptoms, physical signs and laboratory values suggestive of systemic disorders including renal, hepatic, blood, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, and other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteers
* Any medical, social condition, or occupational reason that, in the judgment of the investigator, is a contraindication to protocol participation or impairs the volunteer's ability to give informed consent, increases the risk to the volunteer because of participation in the study, affects the ability of the volunteer to participate in the study or impairs the quality, consistency or interpretation of the study data
* History of non-febrile seizures or atypical febrile seizures

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Incidence and type of Adverse Events | Day of first immunization until one year
  Incidence and type of adverse events (including breakthrough infections), vital signs, clinical laboratory assessments, physical examination findings post first immunization onwards.
  1. Occurrence of solicited symptoms during a 7-day surveillance period after vaccination (day of vaccination (Vx) and +7 days post vaccination)
  2. Occurrence of unsolicited symptoms during a 28-day surveillance period after each vaccination.
  3. Occurrence of serious adverse events during the study period.
  4. Occurrence of Pf infection of vaccine type detected at any point after the first vaccination (retrospectively determined).

SECONDARY OUTCOMES:
Level of Antibodies against Pf proteins in volunteer sera | Post first immunization uptil 56 days post-CHMI or 56 days post-3rd immunization
  1. Antibody titres to pre-erythrocytic stage and erythrocytic stage antigens[PfCSP, PfLSA-1, PfEBA-175 , PfMSP-1, PfMSP-5, EXP-1] by ELISA
  2. Antibody titres to Pf sporozoites, asexual and sexual erythrocytic stage parasites by IFA.
  3. Analysis of antibodies to proteins in the Pf proteome array chip.
Inhibitory Capacity of Volunteer Sera against in vitro Sporozoite Invasion of Hepatocytes | Post first immunization uptil 56 days post-CHMI or 56 days post-3rd immunization
  Capacity of sera from immunized volunteers to inhibit sporozoite invasion (ISI) of hepatocytes in vitro by ISI assay
Quantitation of cellular immune responses against Pf proteins in volunteers | Post first immunization uptil 56 days post-CHMI or 56 days post-3rd immunization
  1. Identification of number of vaccine induced PBMCs following Intracellular cytokine staining by flow cytometry after stimulation with PfSPZ or Pf-infected erythrocytes, peptide pools and P. falciparum infected primary human hepatocyte cell lines.
  2. Identification of numbers of vaccine induced CD4 and CD8 T cells following FluoroSpot assay after stimulation with PfSPZ or Pf-infected erythrocytes.
Whole genome expression profiles of volunteer | Post first immunization uptil 56 days post-CHMI or 56 days post-3rd immunization
  Human gene expression profiling focusing on immune response genes in volunteers

OTHER OUTCOMES:
Time to P. falciparum parasitemia by microscopy over a period of 28 days following CHMI using PfSPZ Challenge by DVI in young adults (aged 18 to 35 years). | Day of CHMI to 28 days later
Proportion of volunteers who develop P. falciparum parasitemia by microscopy over a period of 28 days following CHMI using PfSPZ Challenge by DVI in young adults (aged 18 to 35 years). | Day of CHMI to 28 days later
Time to P. falciparum parasitemia by qPCR over a period of 28 days following CHMI using PfSPZ Challenge by DVI in young adults (aged 18 to 35 years). | Day of CHMI to 28 days later
Proportion of volunteers who develop P. falciparum parasitemia by qPCR over a period of 28 days following CHMI using PfSPZ Challenge by DVI in young adults (aged 18 to 35 years). | Day of CHMI to 28 days later

CONTACTS AND LOCATIONS:
Overall Officials: Salim Abdulla, MD, PHD, Study Director — Ifakara Health Institute (IHI)
Locations (1):
- La Paz Medical Center, Malabo, Equatorial Guinea

REFERENCES:
- [Derived] Jongo SA, Urbano Nsue Ndong Nchama V, Church LWP, Olotu A, Manock SR, Schindler T, Mtoro A, Kc N, Devinsky O, Zan E, Hamad A, Nyakarungu E, Mpina M, Deal A, Bijeri JR, Ondo Mangue ME, Ntutumu Pasialo BE, Nguema GN, Rivas MR, Chemba M, Ramadhani KK, James ER, Stabler TC, Abebe Y, Riyahi P, Saverino ES, Sax J, Hosch S, Tumbo A, Gondwe L, Segura JL, Falla CC, Phiri WP, Hergott DEB, Garcia GA, Maas C, Murshedkar T, Billingsley PF, Tanner M, Ayekaba MO, Sim BKL, Daubenberger C, Richie TL, Abdulla S, Hoffman SL. Safety and Immunogenicity of Radiation-Attenuated PfSPZ Vaccine in Equatoguinean Infants, Children, and Adults. Am J Trop Med Hyg. 2023 May 9;109(1):138-146. doi: 10.4269/ajtmh.22-0773. Print 2023 Jul 5. PMID 37160281